CLINICAL TRIAL: NCT02533167
Title: Impact of Skin to Skin Contact on Maternal Satisfaction, Pain Scores, and Narcotic Usage After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00033101
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Skin to Skin Contact in Cesarean Deliveries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- skin to skin (Experimental): skin to skin initiated on all consented CS while in the operating room
  Interventions: Other: skin to skin

INTERVENTIONS:
Other: skin to skin — initiating skin to skin is not currently the standard of care at our facility so there is 1 interventional arm for this study. control group of no skin to skin until recovery room already established as is the standard of care.

SUMMARY:
Early skin to skin contact has beneficial effects and is part of the Healthy Birth Initiative. Positive effects on breast feeding, cardiorespiratory status, blood glucose control, and temperature has been demonstrated. It is the standard of care for vaginal deliveries but surgery is a barrier in its initiation in the operating room. This study is evaluating initiating skin to skin contact as soon as feasible in the operating room. Informed consent will be obtained from scheduled/non emergent cesarean sections who are of EGA.37 weeks who are ASA I-II and receiving the standard spinal anesthetic. Skin to skin contact will be initiated after delivery as soon as apgars and newborn assessment has been completed. Goal is a minimum of 60 minutes of skin to skin contact between the mother and the newborn, with the only interruption being upon movement from the OR table to the stretcher when leaving the OR. Subjects seen post delivery day 1 for assessments of pain and maternal satisfaction utilizing a sliding 100mm VAS assessment tool.

DETAILED DESCRIPTION:
Initiation of skin to skin contact between the mother and the baby will be done in the operating room during surgery rather than waiting until the recovery room as is our standard of care. After assurance that both mom and newborn are stable, the newborn will be placed across the mother's chest and covered with a blanket to help maintain body temperature. The skin to skin contact is maintained throughout the remaining surgical time and then continued into the recovery room. The subjects are seen post delivery day 1 for evaluation of their pain and satisfaction with care using a 0-100mm sliding VAS scale, with 0=not satisfied at all or no pain at all through 100 = total satisfaction and most severe pain ever.

ELIGIBILITY:
Inclusion Criteria:

* non emergent cesarean deliveries term gestation age ASA I or II spinal anesthetic

Exclusion Criteria:

* contraindication to spinal anesthetic or to medications utilized emergence cesarean delivery under age 18 less than 37 weeks gestational age

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Tonidandel, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Novant Health Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were approached in the preoperative holding room area regarding participation in this study. Subjects were electively scheduled to have a cesarean delivery with proposed healthy outcomes with term deliveries.
Period: Overall Study
Arm/Group | Skin to Skin
Started | 70
Completed | 55
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Maternal Evoked Pain Scores
Description: maternal evoked pain is evaluated utilizing a 100 mm Sliding VAS scale with 0=no pain through 100=most severe pain ever
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
units on a scale | 43.55 (25.34)

2. Other Pre Specified Outcome: Morphine Usage
Description: 24 hour morphine equivalents required in the operating room up to the initial 24 hours after delivery for pain management
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: mg of morphine
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
mg of morphine | 21.83 (19.78)

3. Other Pre Specified Outcome: Maternal Satisfaction With Anesthesia Care
Description: maternal satisfaction with anesthesia care will be evaluated on post delivery day 1 utilizing a 100mm sliding scale where VAS 0= not satisfied at all up to 100= extremely satisfied
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
units on a scale | 95.91 (8.19)

4. Other Pre Specified Outcome: Maternal Satisfaction With Pain Control in the Operating Room
Description: with pain control in the operating room will be evaluated on post delivery day 1 utilizing a 100mm sliding scale VAS 0= not satisfied at all up to 100= extremely satisfied
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
units on a scale | 94.93 (15.52)

5. Other Pre Specified Outcome: Maternal Satisfaction With Postoperative Pain Control
Description: with pain control at 24 hours postoperative will be evaluated on post delivery day 1 utilizing a 100mm sliding scale VAS 0= not satisfied at all up to 100= extremely satisfied
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Skin to Skin: skin to skin initiated on all consented CS while in the operating room
  skin to skin: initiating skin to skin in the operating room
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
units on a scale | 81.52 (23.68)

6. Other Pre Specified Outcome: Maternal Satisfaction-operating Room
Description: maternal satisfaction with operating room atmosphere will be evaluated on post delivery day 1 utilizing a 100mm sliding scale VAS 0= not satisfied at all up to 100= extremely satisfied
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Skin to Skin
Number analyzed (Participants) | 55
units on a scale | 95.98 (8.94)

ADVERSE EVENTS:
Time Frame: 24 hours evaluation time period
Arm/Group | Skin to Skin
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes